CLINICAL TRIAL: NCT02575456
Title: A Single-Center, Randomized, Blind, Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of the Adenovirus Type 5 Vector Based Ebola Virus Disease Vaccine (Ad5-EBOV) in Healthy Adults in Sierra Leone
Brief Title: A Clinical Trial to Evaluate the Recombinant Human Type5 Adenovirus Vector Based Ebola Virus Disease Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Beijing Institute of Biotechnology (Other); Tianjin Cansino Biotechnology Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT024
Record Dates: First submitted 2015-10-11; First posted 2015-10-14 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2015-12

CONDITIONS: Ebola Disease
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Ebola Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): (4×10^10vp/vial, 4 vials): 1 ml sterilization injection water per dose to dilute 2 vials (4×10^10 vp/vial), one shot in each arm, total dose of 1.6×10^11vp. The inoculation site was the central lateral deltoid in the upper arm, and inoculation route was intramuscular injection
  Interventions: Biological: Ebola Vaccine
- Group B (Experimental): (4×10^10vp/vial, 2 vials): 1 ml sterilization injection water per dose to dilute 1 vial (4×10^10vp/vial), total dose of 8×10^10vp, one shot in each arm. The inoculation site was the central lateral deltoid in the upper arm, and inoculation route was intramuscular injection
  Interventions: Biological: Ebola Vaccine
- Group C (Placebo Comparator): (0 vp/ vial, 2 vials):1 ml sterilization injection water per dose to dilute 1 vial, total dose of 0 vp. The inoculation site was the central lateral deltoid in the upper arm, and inoculation route was intramuscular injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ebola Vaccine
  Arms: Group A; Group B
Biological: Placebo — control
  Arms: Group C

SUMMARY:
A Single-Center, Randomized, Blind, Phase II Clinical Trial to Evaluate the Safety and Immunogenicity of the Adenovirus Type 5 Vector Based Ebola Virus Disease Vaccine (Ad5-EBOV) in Healthy Adults Aged Between 18 and 50 years in Sierra Leone.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50 years
* Able to understand the content of informed consent and signed the informed consent
* Able and willing to complete all the secluded study process during the whole study follow-up period (about 6 months).
* Negative in HIV diagnostic blood test on day of enrollment
* Axillary temperature ≤37.0°C on the day of enrollment
* Non-pregnant females with a negative result in the urine pregnancy test on day of enrollment
* General good health as established by medical history and physical examination.

Exclusion Criteria:

* Infected by Ebola virus (inquiry)
* Vaccination with other Ebola vaccine (inquiry)
* HIV infection or other serious immunodeficiency disease (inquiry)
* Allergic history of any vaccination or drugs, or allergic to any ingredient of the Ad5-EBOV, such as mannitol
* Family history of brain or mental disease
* Woman who is pregnant or breast-feeding
* Any acute fever disease or infections in last 7 days
* Major congenital defects or not well-controlled chronic illness
* Asplenia or functional asplenia
* Platelet disorder or other bleeding disorder
* Faint at the sight of blood or needles.
* Prior administration of immunodepressant or corticosteroids, antianaphylaxis treatment, cytotoxic treatment in last 6 months
* Prior administration of other research medicines in last 1 month
* Prior administration of attenuated vaccine(s) in the last one month
* Prior administration of inactivated vaccine(s) in the last 14 days
* Any condition that in the opinion of the investigators may interfere with the participants' compliance or evaluation of study objectives

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of solicited adverse reactions after vaccination | 7 days after vaccination
ELISA antigen-specific assays for antibody to GP responses | 14 days after vaccination
ELISA antigen-specific assays for antibody to GP responses | 28 days after vaccination
ELISA antigen-specific assays for antibody to GP responses | 168 days after vaccination

SECONDARY OUTCOMES:
Occurrence of unsolicited adverse reactions after vaccination | 28 days after vaccination
Occurrence of serious adverse reaction during the whole follow-up period | 6 months
Post-vaccination Rate of infected with HIV | 6 months
Neutralizing antibody titers response to human Ad5 | 14 days after vaccination
Neutralizing antibody titers response to human Ad5 | 28 days after vaccination
Neutralizing antibody titers response to human Ad5 | 168 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Alie H Wurie, Principal Investigator — Ministry of Health & Sanitation
Locations (1):
- Dr. Alie H Wurie, Freetown, Sierra Leone